CLINICAL TRIAL: NCT00660660
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Efficacy Study Comparing 4 Weeks of Treatment With Esomeprazole 20 mg qd to Placebo qd in Patients With Heartburn and Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD)
Brief Title: Local Phase IV, Gastroesophageal Reflux Disease (GERD) Sleep Study US
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9612L00122
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; Esophageal Reflux; Gastro-Esophageal Reflux; Regurgitation; Gastric
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nexium 20mg (Experimental): Nexium 20 mg administered once daily as 22.3 mg of esomeprazole magnesium hydrate
  Interventions: Drug: Esomeprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — Nexium 20 mg administered once daily as 22.3 mg of esomeprazole magnesium hydrate
  Other Names: Nexium
  Arms: Nexium 20mg
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
The purpose of this research study is to compare the safety and effectiveness (how well the medicine works) of esomeprazole (study drug) to placebo (a capsule that does not contain any medication) taken daily in relieving nighttime heartburn and problems sleeping in patients with gastroesophageal reflux disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

* Prior to the run-in period, a history of heartburn or acid regurgitation for 3 months or longer or any history of EE;
* Prior to the run-in period, nighttime heartburn averaging at least 2 or 3 times per week;
* Prior to the run-in period, a history of sleep disturbances associated with GERD for 1 month or more;

Exclusion Criteria:

* Any condition other than GERD that is either the primary cause of, or a significant contributor to, the patient's sleep disturbance
* Sleep medication (including over-the-counter), antihistamine, benzodiazepine, or anti-anxiety medication use that has not been stable (either in dose or regularity) for at least 3 months or is not expected to remain stable during the patient's participation in the study. Patients on a stable regimen, whose regimen is also expected to remain stable throughout the study, are eligible for participation;
* Proton Pump Inhibitor (PPI) use within 1 week prior to Screening. The only allowable acid modifying rescue medication is GELUSIL® during the run-in period. Only study medication and rescue medication (GELUSIL®) is allowed during the treatment period for treatment of acid mediated symptoms

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tore Lind, MD, Study Director — AstraZeneca; Kurt Brown, MD, Study Director — AstraZeneca; David Johnson, MD, Principal Investigator — Eastern Virginia Medical School
Locations (45):
- United States (45):
  - Research Site, Huntsville, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Burbank, California
  - Research Site, Castro Valley, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, DeLand, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, South Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Stockbridge, Georgia
  - Research Site, Overland Park, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Hollywood, Maryland
  - Research Site, Las Vegas, Nevada
  - Research Site, Medford, New Jersey
  - Research Site, Perth Amboy, New Jersey
  - Research Site, West Orange, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Binghamton, New York
  - Research Site, Huntersville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Chattanooga, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Fort Worth Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Ogden, Utah
  - Research Site, Burke, Virginia
  - Research Site, Christiansburg, Virginia
  - Research Site, Fredericksburg, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Bellevue, Washington

REFERENCES:
- [Derived] Johnson DA, Le Moigne A, Hugo V, Nagy P. Rapid resolution of sleep disturbances related to frequent reflux: effect of esomeprazole 20 mg in two randomized, double-blind, controlled trials. Curr Med Res Opin. 2015 Feb;31(2):243-50. doi: 10.1185/03007995.2014.991818. Epub 2015 Jan 9. PMID 25478944
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=437&filename=CSR-D9612L00122.pdf
- See also: CSR-D9612L00122.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=437&filename=CSR-D9612L00122.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The baseline figures shown will be for the modified intention to treat population.
  One patient in each treatment group did not receive study drug; therefore, the safety population has one less patient in each treatment than does the randomized study population.
Groups:
- Nexium 20 mg: Nexium 20 mg administered once daily as 22.3 mg of esomeprazole magnesium hydrate
- Placebo: Capsule once daily (QD)
Period: Overall Study
Arm/Group | Nexium 20 mg | Placebo
Started | 143 (Randomized) | 133 (Randomized)
Met Criteria for MITT Population | 137 | 125
Completed | 138 (Number of completed patients is based on randomized population (143) minus withdrawals (5).) | 124 (Number of completed patients is based on randomized population (133) minus withdrawals (9).)
Not Completed | 5 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 6
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Incorrect enrollment and other | 0 | 1
Not completed — New medication after randomization | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nexium 20 mg | Placebo | Total
Number analyzed (Participants) | 137 | 125 | 262
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.0 (11.7) | 46.8 (12.9) | 46.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 85 | 174
  Male | 48 | 40 | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Relief of Nighttime Heartburn During the Last 7 Days of the Study.
Description: Relief of nighttime heartburn on patient's last 7 days in the study. Relief was defined as a daily diary card response of "none" or 0, on at least 6 of 7 days, allowing for one "mild" or 1 response. Diary card scale (none, mild, moderate, severe).
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 34.3 | 10.4

2. Secondary Outcome: Change in Mean (Average) Pittsburgh Sleep Quality Index (PSQI) Scores From Baseline
Description: To assess the impact of treatment as measured by: Change in global Pittsburgh Sleep Quality Index (PSQI) scores from baseline to week 4. Scale details -'Scoring ranged from 0, "no difficulty" to 3, "severe difficulty." Items were grouped into 7 component scores. The 7 components were then summed to yield a global PSQI score. Global scores >5 were considered to meet the criteria of sleep disturbance.
Time Frame: Baseline and 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 134 | 123
Scores on a scale | -2.93 (0.34) [lower limit 0.3400] | -1.80 (0.34) [lower limit 0.3400]

3. Secondary Outcome: Achievement of Developer-defined Good Sleep
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on sleep disturbances associated with Gastroesophageal reflux disease (GERD), as measured by achievement of (yes/no) developer-defined good sleep (global Pittsburgh Sleep Quality Index - PSQI score ≤5) at Week 4.
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 21 | 29
Participants | 19 | 24

4. Secondary Outcome: Number of Patients With Complete Resolution of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) After 1 Week of Treatment.
Description: The assessment was based on patients registrations of the answers "Yes" or "No" to the question: "Did you have trouble sleeping last night due to your heartburn or other symptoms of Gastroesophageal Reflux Disease (GERD)?". Complete resolution of GERD-related sleep disturbances was defined as a daily diary response of "No" on 7 consecutive days.
Time Frame: 1 week
Measure: Number; unit: Participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Participants | 44 | 23

5. Secondary Outcome: Number of Patients With Complete Resolution of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) After 2 Weeks of Treatment.
Description: The assessment was based on patients registrations of the answers "Yes" or "No" to the question: "Did you have trouble sleeping last night due to your heartburn or other symptoms of Gastroesophageal Reflux Disease (GERD)?". Complete resolution of GERD-related sleep disturbances was defined as a daily diary response of "No" on 14 consecutive days.
Time Frame: 2 weeks
Measure: Number; unit: Participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Participants | 54 | 20

6. Secondary Outcome: Number of Patients With Complete Resolution of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) After 4 Weeks of Treatment.
Description: The assessment was based on patients registrations of the answers "Yes" or "No" to the question: "Did you have trouble sleeping last night due to your heartburn or other symptoms of GERD?". Complete resolution of Gastroesophageal Reflux Disease (GERD)-related sleep disturbances was defined as a daily diary response of "No" on 7 consecutive days during 4 weeks of treatment.
Time Frame: 4 weeks
Measure: Number; unit: Participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Participants | 29 | 14

7. Secondary Outcome: Number of Patients With Complete Resolution of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) on the Patient's Last 7 Days in the Study.
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on sleep disturbances associated with Gastroesophageal Reflux Disease (GERD), as measured by: Complete resolution of sleep disturbances on the patient's last 7 days in the study.
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Participants | 66 | 27

8. Secondary Outcome: Number of Patients With Relief of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) After 1 Week of Treatment
Description: The assessment was based on patients registrations of the answers "Yes" or "No" to the question: "Did you have trouble sleeping last night due to your heartburn or other symptoms of Gastroesophageal Reflux Disease (GERD)?". Relief of sleep disturbances associated with GERD was defined as a daily diary response of "Yes" on not more than 2 of 7 consecutive days.
Time Frame: 1 week
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Participants | 79 | 53

9. Secondary Outcome: Number of Patients With Relief of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) After 2 Weeks of Treatment
Description: as for outcome 8
Time Frame: 2 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Participants | 90 | 54

10. Secondary Outcome: Number of Patients With Relief of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) After 4 Weeks of Treatment
Description: as for outcome 8
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Participants | 74 | 45

11. Secondary Outcome: Percentage of Patients With Relief of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) on the Patient's Last 7 Days in the Study.
Description: as for outcome 8
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of Participants | 71.5 | 55.2

12. Secondary Outcome: Percentage of Days Without Gastroesophageal Reflux Disease (GERD)-Related Sleep Disturbances During the 4 Week Period
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on sleep disturbances associated with Gastroesophageal Reflux Disease (GERD)as measured by: Percent of days without sleep disturbances after 4 weeks of treatment. Each morning of the study, patients registered their answer "Yes" or "No" to the question, "Did you have trouble sleeping last night due to your heartburn or other symptoms of GERD?" in the diary card.'
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 124
Percentage of days | 73.0 (29.7) | 59.3 (29.9)

13. Secondary Outcome: Number of Days to First Relief of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) During the 4 Week Treatment Period
Description: The assessment was based on patients registrations of the answers "Yes" or "No" to the question: "Did you have trouble sleeping last night due to your heartburn or other symptoms of Gastroesophageal Reflux Disease (GERD)?". Relief of sleep disturbances associated with GERD was defined as a daily diary response of "Yes" on not more than 2 of 7 consecutive days, and 'days to first relief' was defined as the first day of the 7 days that reached relief of sleep disturbance.
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Days | 1 [1 to 21] | 3 [1 to 21]

14. Secondary Outcome: Number of Days to Resolution of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) During the 4 Week Treatment Period
Description: as for outcome 8
Time Frame: 4 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Days | 1 [1 to 14] | 2 [1 to 21]

15. Secondary Outcome: Number of Days to First Complete Resolution of Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD) During the 4 Week Treatment Period
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on sleep disturbances associated with Gastroesophageal Reflux Disease (GERD), as measured by: Days to complete resolution of sleep disturbance. Days to complete resolution of sleep disturbances associated with GERD was defined as the number of days until the first day of the first 7-consecutive-day period during which the patient's daily diary response was "No" (did not have trouble sleeping due to GERD symptoms).'
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Days | 9 [1 to 21] | 21 [1 to 21]

16. Secondary Outcome: Percentage of Patients With Complete Resolution of Daytime Heartburn After 1 Week of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of daytime heartburn after 1 week of treatment. Results based on MITT population with available data for this outcome measure. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: 1 week
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 22 | 4

17. Secondary Outcome: Percentage of Patients With Complete Resolution of Daytime Heartburn After 2 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of daytime heartburn after 2 weeks of treatment. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: 2 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 37 | 11

18. Secondary Outcome: Percentage of Patients With Complete Resolution of Daytime Heartburn After 4 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of daytime heartburn after 4 weeks of treatment. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 35 | 7

19. Secondary Outcome: Percentage of Patients With Complete Resolution of Daytime Heartburn on the Patient's Last 7 Days in the Study
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of daytime heartburn on the patient's last 7 days in the study. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 45 | 9

20. Secondary Outcome: Percentage of Patients With Complete Resolution of Nighttime Heartburn After 1 Week of Treatment.
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of nighttime heartburn after 1 week of treatment. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: 1 week
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 23 | 4

21. Secondary Outcome: Percentage of Patients With Complete Resolution of Nighttime Heartburn After 2 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of nighttime heartburn after 2 weeks of treatment. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: 2 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 36 | 6

22. Secondary Outcome: Percentage of Patients With Complete Resolution of Nighttime Heartburn After 4 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of nighttime heartburn after 4 weeks of treatment. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 25 | 6

23. Secondary Outcome: Percentage of Patients With Complete Resolution of Nighttime Heartburn on the Patient's Last 7 Days in the Study.
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of nighttime heartburn on the patient's last 7 days in the study. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 42 | 8

24. Secondary Outcome: Percentage of Patients With Complete Resolution of 24-hour Heartburn After 1 Week of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of 24-hour heartburn after 1 week of treatment. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: 1 week
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 16 | 3

25. Secondary Outcome: Percentage of Patients With Complete Resolution of 24-hour Heartburn After 2 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of 24-hour heartburn after 2 weeks of treatment. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: 2 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 30 | 4

26. Secondary Outcome: Percentage of Patients With Complete Resolution of 24-hour Heartburn After 4 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of 24-hour heartburn after 4 weeks of treatment. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 30 | 4

27. Secondary Outcome: Percentage of Patients With Complete Resolution of 24-hour Heartburn on the Patient's Last 7 Days in the Study
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Complete resolution of 24-hour heartburn on the patient's last 7 days in the study. Complete resolution of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "None" on 7 consecutive days.
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 37 | 5

28. Secondary Outcome: Percentage of Patients With Relief of Daytime Heartburn After 1 Week of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of daytime heartburn after 2 weeks of treatment. Results based on MITT population with available data for this outcome measure. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.'
Time Frame: 1 week
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 34 | 13

29. Secondary Outcome: Percentage of Patients With Relief of Daytime Heartburn After 2 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of daytime heartburn after 2 weeks of treatment. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.'
Time Frame: 2 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 48 | 14

30. Secondary Outcome: Percentage of Patients With Relief of Daytime Heartburn After 4 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of daytime heartburn after 4 weeks of treatment. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.'
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 40 | 9

31. Secondary Outcome: Percentage of Patients With Relief of Daytime Heartburn on the Patient's Last 7 Days in the Study
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of daytime heartburn on the patient's last 7 days in the study. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.'
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 55 | 14

32. Secondary Outcome: Percentage of Patients With Relief of Nighttime Heartburn After 1 Week of Treatment.
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of nighttime heartburn after 1 week of treatment. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.
Time Frame: 1 week
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 28 | 9

33. Secondary Outcome: Percentage of Patients With Relief of Nighttime Heartburn After 2 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of nighttime heartburn after 2 weeks of treatment. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.
Time Frame: 2 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 40 | 7

34. Secondary Outcome: Percentage of Patients With Relief of Nighttime Heartburn After 4 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of nighttime heartburn after 4 weeks of treatment. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 26 | 6

35. Secondary Outcome: Percentage of Patients With Relief of Nighttime Heartburn on the Patient's Last 7 Days in the Study
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of nighttime heartburn on the patient's last 7 days in the study. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 47 | 13

36. Secondary Outcome: Percentage of Patients With Relief of 24-hour Heartburn After 1 Week of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of 24-hour heartburn after 1 week of treatment. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.
Time Frame: 1 week
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 27 | 5

37. Secondary Outcome: Percentage of Patients With Relief of 24-hour Heartburn After 2 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of 24-hour heartburn after 2 weeks of treatment. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.
Time Frame: 2 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 36 | 5

38. Secondary Outcome: Percentage of Patients With Relief of 24-hour Heartburn After 4 Weeks of Treatment
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of 24-hour heartburn after 4 weeks of treatment. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 33 | 5

39. Secondary Outcome: Percentage of Patients With Relief of 24-hour Heartburn on the Patient's Last 7 Days in the Study
Description: To assess the impact of treatment with Esomeprazole 20 (E20) versus placebo on heartburn, as measured by: Relief of 24-hour heartburn on the patient's last 7 days in the study. Relief of daytime, nighttime, and 24-hour heartburn was defined as a daily diary response of "none" on at least 6 of 7 days, allowing for 1 "mild" response.
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 45 | 9

40. Secondary Outcome: Percentage of Patients With Nighttime Heartburn Symptom Improvement From Baseline During the Last 7 Days in the Study
Description: Number and percentage of patients with nighttime heartburn symptom improvement based on weekly symptom scores at Baseline compared to the last week of study drug treatment. Symptom improvement was defined as any decrease in weekly symptom score from Baseline until the last 7 days in the study.
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 89.8 | 83.2

41. Secondary Outcome: Percentage of Participants With Daytime Heartburn Symptom Improvement From Baseline During the Last 7 Days in the Study
Description: Number of patients with daytime heartburn symptom improvement based on weekly symptom scores at Baseline compared to the last week of study drug treatment. Symptom improvement was defined as any decrease in weekly symptom score from Baseline until the last 7 days in the study.
Time Frame: Days 21-28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 137 | 125
Percentage of participants | 86.1 | 76

42. Secondary Outcome: Percentage of Patients With 24-hour Heartburn Symptom Improvement From Baseline During the Last 7 Days in the Study.
Description: Number of patients with 24-hour heartburn symptom improvement based on weekly symptom scores at Baseline compared to the last week of study drug treatment. Symptom improvement was defined as any decrease in weekly symptom score from Baseline until the last 7 days in the study.
Time Frame: Days 21- 28 (for early dropouts the last 7 days staying in the study)
Population: Results based on MITT population with available data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 125 | 137
Percentage of participants | 89.8 | 80

43. Secondary Outcome: Equivalent Number of Hours Lost Because of Sleep Disturbances Due to Gastroesophageal Reflux Disease (GERD) Symptoms (Average)
Time Frame: 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Work hours
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 78 | 74
Work hours | 8.9 (11.1) | 5.2 (11.7)

44. Secondary Outcome: Change From Baseline in Percent of Work Impairment Because of Sleep Disturbances Due to Gastroesophageal Reflux Disease (GERD) Symptoms (Average)
Description: Degree of sleep disturbance affecting work productivity. 100% is considered to be the worst outcome where there is no ability to work. 0% is considered to be the best outcome, no impairment.
Time Frame: Baseline and 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 83 | 78
Percentage | -25.3 (28.7) | -14 (27.4)

45. Secondary Outcome: Change From Baseline in Percent Overall Work Impairment Due to Sleep Disturbance (Average)
Description: Equivalent number of work hours missed was derived from questions 2, 4 and 5 of the Work Productivity and Activity Impairment Questionnaire: Sleep Disturbance-GERD (Gastroesophageal Reflux Disease) and summed up with the percent work impairment during the remaining hours that were actually worked.
Time Frame: Baseline and 4 weeks
Population: Results based on MITT population with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 76 | 74
Percentage | -24.8 (29.5) | -14.9 (25.9)

46. Secondary Outcome: Change From Baseline in Percent Activity Impairment Due to Sleep Disturbances (Average)
Description: as for outcome 2
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 87 | 78
Percentage | -25.1 (27.4) | -17.1 (28)

47. Secondary Outcome: Monetary Value of Work Hours Saved
Description: The monetary value of the work hours saved was derived from questions 2,4, and 5 of the WPAI and a standard hourly compensation rate reported by the US Bureau of Labor Statistics (US$28.48 as of June 2008).
Time Frame: Week 4
Population: Results based on MITT population with available data for this outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: Monetary value (US dollars)
Arm/Group | Nexium 20 mg | Placebo
Number analyzed (Participants) | 76 | 74
Monetary value (US dollars) | 280.21 (34.88) [34.8800 to 0.0000] | 156.61 (33.05) [33.05 to 0.0000]

ADVERSE EVENTS:
Arm/Group | Nexium 20 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/143 | 1/133
Other Adverse Events (participants affected / at risk) | 0/143 | 0/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nexium 20 mg (N=143) | Placebo (N=133)
Pneumonia (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Sponsor does not publish within 2 years after study completion, PI is permitted to publish, with confidential information removed from manuscript. Sponsor will have opportunity to review and approve publication at least 60 days prior to being submitted/disclosed. Sponsor can request, in writing, an additional 90 day embargo.